CLINICAL TRIAL: NCT04137263
Title: A Prospective, Study Evaluating the Efficacy of DOSE Formulations in Treatment of Melasma and Cutaneous Signs of Aging
Brief Title: Study Evaluating the Efficacy of DOSE Formulations in Treating Melasma and Cutaneous Signs of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOSE-2019-01
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2020-12

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Subjects will receive dose formulation for treatment of melasma
  Interventions: Other: DOSE formulation

INTERVENTIONS:
Other: DOSE formulation — over-the-counter topical

SUMMARY:
The primary objective is to evaluate the efficacy, of D.O.S.E formulations in the treatment of melasma and cutaneous signs of aging.

DETAILED DESCRIPTION:
Melasma is a hyperpigmentation disorder that presents as irregularly shaped macules on the face of women. The etiology is unknown however there is strong evidence that genetics, hormones, sun exposure can trigger and worsen the disease. Increased dermal vascularity and expression of angiogenic factors also seem to play a role. Melasma is a chronic and relapsing condition, that is difficult to treat, and can have a negative impact on quality of life.

Numerous treatments exist for melasma including topical lightening agents, chemical peels, and a variety of laser and light based options. Long-term management is difficult as topical agents can often cause irritation, burning, peeling and inflammatory hyperpigmentation. Light based therapies can also lead to relapse or worsening of the disease.

Melasma, in combination with photodamage from cumulative sun exposure and aging, can lead to a complex picture when making a skin care plan for a cosmetic patient. The custom D.O.S.E professional service can be utilized to make a personalized serum to improve skin discoloration and the visible signs of aging. The purpose of this study is to evaluate the efficacy of D.O.S.E formulations in the treatment of melasma and visible signs of aging.

ELIGIBILITY:
Inclusion Criteria:

* 1. Females age 18-65, Fitzpatrick skin types I-VI 2. Mild to moderate melasma 3. Half of subjects with hypervascular melasma identified by Visia complexion analysis 4. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedures.

  5. Willingness to abstain from any other procedures to the areas to be treated throughout the trial period.

  6. Willingness and ability to comply with protocol requirements, including adherence to photography and returning for follow-up visits.

  7. Women of childbearing potential willing to use an acceptable form of birth control during trial period.
  1. Hormonal contraception - pill, injection, implant, patch, vaginal ring, Intrauterine device
  2. Intrauterine coil
  3. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
  4. Abstinence (If practicing abstinence must agree to use barrier method described above (c) if becomes sexually active).
  5. Vasectomized partner (Must agree to use barrier method described above (c) if becomes sexually active with an Un-Vasectomized partner).

     8. Female patients will be either of non-childbearing potential defined as: Having no uterus and/or both ovaries, postmenopausal (no menses for at least 12 months prior), or has had a bilateral tubal ligation at least 6 months prior to study enrollment.

     Exclusion Criteria:
* 1. Pregnancy, currently breast feeding or planning pregnancy for the duration of the trial.

  2. Known hypersensitivity or allergy to the components of the study medication. 3. Concurrent enrollment in any study involving the use of investigational devices or drugs.

  4. Current smoker or history of smoking in the last five years. 5. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.

  6. Presence of an active systemic or local skin disease that may affect treatment area.

  7. History of the following cosmetic treatments to the area(s) to be treated:
  1. Energy based device or laser procedure to the area within the past 6 months (Ultherapy, ablative and non-ablative laser, intense pulsed light, etc)
  2. Medium to deep chemical peels (e.g. TCA, Phenol) for 6 months or light chemical peels (e.g. Glycolic Acid >20%) within the past 3 months; 8. History of using the following cosmetic, OTC or prescription medications:

  a. Topical glycolic acid (5% or greater) in the past 4 weeks. b. Topical or oral tranexamic acid within in the past 4 weeks (e.g. Lytera 2.0); c. Topical Retinoids (e.g. Rx tretinoin or OTC retinol) within the past four weeks; d. Topical hydroquinone within the past 4 weeks; e. Topical salicylic acid within the past 4 weeks; f. Topical or oral corticosteroids within the past 4 weeks; g. Other topical products intended to treat melasma within the past 4 weeks; 9. Individuals who started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to study entry or who plan on starting, stopping, or changing doses of HRT or hormones for birth control during the study.

  10. Any planned surgical intervention to the treatment area for the duration of the trial 11. Any visible surface alteration to the treatment area that may interfere with evaluation, at investigator discretion 12. Any pre-existing medical condition that may interfere with study compliance or evaluation, at investigator discretion 13. Inability to comply with all study protocols and regulations 14. Current taking an immunosuppressant or applying a topical corticosteroid to the affected area

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Improvement of Melasma | Baseline to Day 120
  change in Investigator MoPASI score

CONTACTS AND LOCATIONS:
Overall Officials: Monica Boen, M.D., Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No